CLINICAL TRIAL: NCT01617902
Title: Hyperbilirubinemia After Major Cardiac or Thoracic Aorta Surgery: Predictors and Clinical Significance
Brief Title: Hyperbilirubinemia After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joon Bum Kim, Assistant Professor, Asan Medical Center
Other Study IDs: HBCS_01
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Diseases
Keywords: Hyperbilirubinemia; cardiac; surgery; aorta; prognosis
MeSH Terms: conditions — Cardiovascular Diseases; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to evaluate the incidence and risk factors of hyperbilirubinemia following major cardiac or thoracic aorta surgery, and to determine the clinical impacts of the hyperbilirubinemia on postoperative mortality and morbidity.

DETAILED DESCRIPTION:
Patients receiving elective cardiac or thoracic aorta surgery will be monitored for the development of postoperative hyperbilirubinemia. Collection of data will include patient baseline demographic characteristics, laboratory and echocardiographic findings, procedural factors of the surgery, and early postoperative variables. Serial postoperative liver function testings will be done during the hospitalization. Postoperative hyperbilirubinemia is defined as serum bilirubin level of 3mg/dL.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years who are scheduled to undergo elective major cardiac or thoracic aorta surgery. Major cardiac surgery includes coronary artery bypass grafting, pericardiectomy and corrections of cardiac diseases using cardiopulmonary bypassing (valve surgery, tumor excision, arrhythmia surgery, heart transplantation, ventricular reconstruction, pulmonary thromboembolectomy, and atrial or ventricular septal defects closure).

Exclusion Criteria:

1. univentricular or one-and-half ventricle repairs
2. presence of known liver cirrhosis or hepatic cancer
3. history of liver transplantation
4. Genetic diseases that affects bilirubin metabolism (i.e. Gilbert syndrome)
5. preoperative bilirubin level of 3mg/dL or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major cardiac or thoracic aorta surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
All cause-death | Within 30 days after surgery or during postoperative hospitalization

SECONDARY OUTCOMES:
gastrointestinal or hepatobiliary complications requiring intervention | Within 30 days after surgery or during postoperative hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Joon Bum Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea